CLINICAL TRIAL: NCT00095810
Title: An Open-Label Study of Aripiprazole to Evaluate the Safety and Tolerability in Patients With Psychosis Associated With Parkinson's Disease
Brief Title: Aripiprazole in Patients With Psychosis Associated With Parkinson's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka America Pharmaceutical (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CN138-060
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2010-12

CONDITIONS: Parkinson's Disease; Psychoses
Keywords: Psychosis, Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease; Psychotic Disorders | interventions — Aripiprazole

ARMS (1):
- A (Experimental)
  Interventions: Drug: aripiprazole

INTERVENTIONS:
Drug: aripiprazole — Tablets, Oral, 1-10mg, Once daily, 6 weeks.
  Other Names: Abilify

SUMMARY:
The purpose of this clinical research study is to assess the safety and tolerability of aripiprazole in patients with psychosis associated with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of idiopathic Parkinson's disease.
* Psychosis related to Parkinson's disease.

Exclusion Criteria:

* Psychosis present prior to diagnosis of Parkinson's disease.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2003-07; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Tolerability

SECONDARY OUTCOMES:
Safety Assessments

CONTACTS AND LOCATIONS:
Locations (1):
- Local Institution, Albany, New York, United States

REFERENCES:
- [Background] Friedman JH, Berman RM, Goetz CG, Factor SA, Ondo WG, Wojcieszek J, Carson WH, Marcus RN. Open-label flexible-dose pilot study to evaluate the safety and tolerability of aripiprazole in patients with psychosis associated with Parkinson's disease. Mov Disord. 2006 Dec;21(12):2078-81. doi: 10.1002/mds.21091. PMID 17013906
- See also: PhRMA website-CSR Synopsis — http://www.ncbi.nlm.nih.gov/pubmed/17013906?dopt=Abstract